CLINICAL TRIAL: NCT04657029
Title: The Acute Effects of Aerobic Exercise on Sensorimotor Adaptation in Chronic Stroke
Brief Title: Aerobic Exercise and Sensorimotor Adaptation in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ChrisMackaySensMotStroke2020
Record Dates: First submitted 2020-11-22; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Stroke
Keywords: sensorimotor adaptation; aerobic exercise
MeSH Terms: conditions — Stroke | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: In a cross-over design, each participant was pseudo-randomised to complete an intervention condition (Treadmill) or control condition (Rest) first, returning at least one week later (washout period) to complete the alternate condition. A minimum washout period of one week was used to allow for any physiological changes due to exercise to return to resting levels, but to minimise any stroke recovery-associated changes to function. Participants were asked to refrain from exercising in the 24 hours prior to their visit. At each visit, participants completed the sensorimotor adaptation task on two occasions, pre and post intervention, resulting in four assessment timepoints (PreControl, PostControl and PreTreadmill, PostTreadmill). The post intervention assessment aimed to commence within 15 minutes of completing the treadmill or rest condition.
Who Masked: Outcomes Assessor
Masking Description: Blinded Assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill condition (Experimental): The intervention condition consisted of a single session of moderate-high intensity aerobic exercise (65% of heart rate reserve) for 30 minutes walking on a standard treadmill. The single treadmill session included a progressive increase in intensity to reach the target heart rate (approx. 5 mins) as well as a cooling down period (approx. 5 mins). The warm-up and cool-down were included as part of the total 30 minutes of walking exercise. Target heart rates were calculated using the Karvonen method [25] with levels adjusted for those taking heart rate lowering medications (i.e. beta blockers), following methods previously published in post stroke populations [26, 27]. Participants were asked to self-rate their intensity of exercise every 10 minutes verbally using BORG's 6-20 scale rating of perceived exertion [28]. Participants were instructed to walk at a pace that resulted in a rating between 11 (fairly light) and 14 (somewhat hard) on the scale.
  Interventions: Behavioral: Treadmill
- Control condition (Other): The control condition involved an equivalent time period (30 minutes) of seated resting where participants were provided with an education session about the impact and effects of stroke by the same research assistant.
  Interventions: Behavioral: Treadmill

INTERVENTIONS:
Behavioral: Treadmill — 30 minutes of moderate-high intensity treadmill training.

SUMMARY:
A single-blinded crossover study. Participants attended two separate sessions at the university campus, completing an aerobic exercise intervention in one session and a resting control condition in the other session. Sensorimotor adaptation was assessed before and after each session. Participants were twenty people with chronic stroke. Intervention completed was treadmill exercise at mod-high intensity for 30 minutes.

DETAILED DESCRIPTION:
Participants Twenty people with chronic stroke participated in the study (aged 61 ± 13 years; 76% male).

Experimental design In a cross-over design, each participant was pseudo-randomised to complete an intervention condition (Treadmill) or control condition (Rest) first, returning at least one week later (washout period) to complete the alternate condition. A minimum washout period of one week was used to allow for any physiological changes due to exercise to return to resting levels, but to minimise any stroke recovery-associated changes to function. Participants were asked to refrain from exercising in the 24 hours prior to their visit. At each visit, participants completed the sensorimotor adaptation task on two occasions, pre and post intervention, resulting in four assessment timepoints (PreControl, PostControl and PreTreadmill, PostTreadmill). The post intervention assessment aimed to commence within 15 minutes of completing the treadmill or rest condition.

Intervention The intervention condition consisted of a single session of moderate-high intensity aerobic exercise (65% of heart rate reserve) for 30 minutes walking on a standard treadmill (Landice L7 treadmill), with arms placed comfortably by participants on the rail (in front) or swinging freely. Information describing the specific features of the training session (e.g. heart rate, blood pressure response, treadmill speed, total distance walked) were recorded to monitor the response to exercise and adherence to the exercise protocol. The single treadmill session included a progressive increase in intensity (usually increased speed, or gradient) to reach the target heart rate (approx. 5 mins) as well as a cooling down period (approx. 5 mins) to allow for participants to return towards resting levels for vital observations. The warm-up and cool-down were included as part of the total 30 minutes of walking exercise. Target heart rates were calculated using the Karvonen method with levels adjusted for those taking heart rate lowering medications (i.e. beta blockers), following methods previously published in post stroke populations. Heart rate was measured using a chest strap monitor (polar-electro) and monitored by a research assistant who facilitated changes in treadmill parameters to enable participants to reach their target. Participants were asked to self-rate their intensity of exercise every 10 minutes verbally using BORG's 6-20 scale rating of perceived exertion. Participants were instructed to walk at a pace that resulted in a rating between 11 (fairly light) and 14 (somewhat hard) on the scale. The control condition involved an equivalent time period (30 minutes) of seated resting where participants were provided with an education session about the impact and effects of stroke by the same research assistant.

Sensorimotor adaptation task Apparatus and setup. Participants were seated in front of a desk (approximately 50 cm from their coronal plane) and asked to move a digitising pen (15.95 cm long, 1.4 cm wide, 17 g) on a digitizing tablet (WACOM Intuos4 PTK 1240, size: 19.2 x 12 in., resolution = 0.25 mm) from an origin to a target point. The pen's position on the tablet (XY coordinates) was sampled at 100 Hz and displayed in real time as a circular cursor with a 5-pixel radius (1.25 mm) on a horizontally placed computer monitor. Direct vision of the hand was prevented by placing the tablet and the hand directly beneath an opaque stand, with the horizontal monitor placed atop the stand.

Task instructions. Participants first received task instructions to move an on-screen cursor from the start to the target, in a straight line, in a single movement, as quickly and as accurately as possible. Further, participants were instructed that the feedback of the movement would be changed from time-to-time, and that participants were to change their movement in response to this change of feedback, whilst keeping movements as straight as possible.

In each trial, the participants' task was to move from the origin location through the target location as quickly and accurately as possible using their dominant upper limb. Targets were presented in one of three locations (210, 225 or 240 degrees from the right horizontal plane) in random order. These target directions were selected such that target-reaching movements involved the horizontal adductors of the shoulder joint. After moving through the target, or past the target, a high-pitched tone sounded to indicate trial completion. Following completion of a trial the origin location was re-displayed immediately and participant directed to repeat task. If the participant did not complete a successful trial, they were directed to return to the origin location and repeat the trial.

First, participants encountered 18 baseline trials under normal (correct) feedback with no rotation. Participants then immediately completed 66 adaptation trials, where the visual feedback on the display monitor was perturbed by rotating it 30 degrees in a clockwise direction (1st testing day) or counter-clockwise direction (2nd testing day). After the adaptation block, to notify participants that the perturbation had been removed, a popup dialog box appeared with the statement "In the next few trials, the disturbance that the computer applied would be removed. Please aim straight to the target." The instructions on-screen were read out by the experimenter to ensure it was understood. This was immediately followed by 6 no-feedback trials. Finally, participants completed 36 washout trials under normal cursor feedback conditions (i.e., no cursor rotation), to return behaviour to an unadapted state.

Data Processing and Analysis Custom scripts written in LabVIEW scored reach directions, which were quantified at the 15th data point (150 milliseconds into the reach), as online movement corrections typically occur after 150 ms into a reach. Trials with reach direction outside a 120 degree range of the target (60 degrees on either side of the target) were discarded as outliers. Trials were binned into cycles of one visit to each of the three targets. The dependent variable was percent adaptation, which quantified reach directions in every cycle relative to the ideal reach direction by calculating reach directions as a percentage of ideal reach directions resulting from perfect adaptation performance. Ideal reach direction was 30 degree clockwise for a 30 degree counter-clockwise rotation, and 30 degrees counter-clockwise for a 30 degree clockwise rotation.

Percent adaptation=100% × (reach direction)/(ideal reach direction)

As observed previously, there was a rapid error reduction phase of reaching where a majority of learning occurred followed by a slower rate of adaptation. Here, as the targets were spaced close together, rapid error reduction occurred in trials 1-9 (i.e., the first three cycles), similar to recent work. At completion of the fourth cycle, adaptation was greater than 70% both before and after the treadmill and control conditions. We thus selected the first three cycles to quantify rapid error reduction.

Individual differences in reach directions at baseline can affect measures of adaptation. Previous methods of accounting for this by subtracting pre-perturbation behaviour from post-perturbation behaviour is more sensitive to noisy baselines and risk of Type 2 error. To account for pre-perturbation baseline biases, we entered percent adaptation averaged from the final three cycles before rotation onset (i.e., percent adaptation in the last five baseline cycles) as covariates in all of our analysis of covariance analyses.

After the adaptation trials, there were two cycles where no feedback was provided to the participant. That is, unlike all previous trials where participants could follow a tracking cursor with their vision, the participants received no real time feedback about where they were reaching. The first no-feedback cycle was taken as a measure of implicit learning, similar to previous work.

Our outcome measures of interest were (1) adaptation performance (2) implicit aftereffects, quantified as reaches that remained adapted despite notification of perturbation removal in the no-feedback block and (3) explicit learning, estimated as the volitional disengagement of adapted behaviour after receiving notification of perturbation removal (i.e., the change in percent adaptation from the mean of the last three adaptation cycles to the first no-feedback cycle after receiving notification that the perturbation was gone), and (4) de-adaptation performance. To evaluate these measures, we ran ANCOVAs with the between-subjects factor Intervention Order (Control First, Treadmill First) and the within-subjects factors: Intervention (Control, Treadmill), Time (Pre-Intervention, Post-Intervention) and (where applicable) Cycles (cycles 1..3), with pre-rotation biases as covariates of no interest (estimated from mean percent adaptation in the last three baseline cycles). Where appropriate, Greenhouse-Geisser corrections were applied. Alpha was set at 0.05. SPSS v24.0 was used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Time of stroke greater than three months ago
* Be able to walk with or without and aid for at least 10 metres
* Understand three stage commands

Exclusion Criteria:

* Unable to walk independently prior to current stroke
* Have co-morbidities that limit their walking (e.g. arthritis, orthopaedic surgery)
* Unstable cardiac status
* Unable to understand three stage commands
* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Sensorimotor adaptation change | Pre and Post intervention and Pre and Post Control. There was one week between the two conditions
  Participants were seated in front of a desk and asked to move a digitising pen on a digitizing tablet from an origin to a target point. The pen's position on the tablet (XY coordinates) was sampled at 100 Hz and displayed in real time as a circular cursor with a 5-pixel radius (1.25 mm) on a horizontally placed computer monitor. Direct vision of the hand was prevented by placing the tablet and the hand directly beneath an opaque stand, with the horizontal monitor placed atop the stand.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neva JL, Ma JA, Orsholits D, Boisgontier MP, Boyd LA. The effects of acute exercise on visuomotor adaptation, learning, and inter-limb transfer. Exp Brain Res. 2019 Apr;237(4):1109-1127. doi: 10.1007/s00221-019-05491-5. Epub 2019 Feb 18. PMID 30778618

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04657029/Prot_SAP_000.pdf